CLINICAL TRIAL: NCT00195390
Title: Investigation of Prevenar (Pneumococcal 7-Valent Conjugate Vaccine) Administration for Post-Marketing Surveillance
Brief Title: Study Investigating Administration of Prevenar for Post-Marketing Surveillance
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 0887X-101583
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Pneumococcal Infections
Keywords: Vaccine; heptavalent pneumococcal conjugate vaccine
MeSH Terms: conditions — Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Biological: Prevenar — Prevenar 0.5ml/ Vial and PFS

SUMMARY:
The purpose of this study is to identify the following problems and questions with respect to the safety of Pneumococcal 7-Valent Conjugate Vaccine (Diphtheria CRM 197 Protein), Prevenar, during the post-marketing period in Korea, as required by Korea Food and Drug Administration (KFDA) regulations.

1. Adverse reactions (especially serious adverse reactions)
2. Incidences of adverse reactions under routine vaccine use
3. Factors that may affect the safety of the vaccine

ELIGIBILITY:
Inclusion Criteria:

* Infants and children aged 6 weeks to 9 years, provided the conditions pertaining to contraindications, warnings, precautions, and interactions stated in the package insert do not apply.

Exclusion Criteria:

* Hypersensitivity to latex or to any component of the vaccine, including diphtheria toxoid
* Suffering from a current or recent febrile illness.

Ages: 6 Weeks to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary care clinic, secondary and tertiary medical centers
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2004-07; Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Seoul, South Korea